CLINICAL TRIAL: NCT01856504
Title: Validation of an Intracycle CT Motion CORrection Algorithm for Diagnostic AccuracY: A Prospective Multicenter Study
Brief Title: Validation of an Intracycle CT Motion CORrection Algorithm for Diagnostic AccuracY
Acronym: VICTORY
Status: Completed | Type: Observational
Sponsor: MDDX LLC (Industry)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: VICTORY
Record Dates: First submitted 2013-05-15; First posted 2013-05-17 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Artery Disease; Coronary Arteriosclerosis
Keywords: Heart Disease; Coronary Artery Disease; Coronary Arteriosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CCTA Patient: 1. Consenting adult patients ≥18 years of age;
  2. Suspected but without known prior history of CAD
  3. Not actively taking heart rate lowering agents at least 48 hours prior to study (e.g., AV nodal blockers such as beta blockers, calcium channel blockers or digoxin)
  4. Glomerular filtration rate >60 ml/min
  5. CCTA and ICA within 1 week of each other with no interscan event (e.g., myocardial infarction or coronary revascularization)

SUMMARY:
To demonstrate the incremental utility of SSF for individuals undergoing CCTA, with expected improvements in image quality and diagnostic accuracy.

DETAILED DESCRIPTION:
Hypothesis: Coronary CT angiography (CCTA) employing a novel intracycle motion compensation algorithm (SnapShot Freeze [SSF]) will be superior to CCTA without an intracycle motion compensation algorithm ("conventional" CCTA) for diagnostic accuracy and image quality.

Scientific Basis: Preliminary study (Leipsic, Min, Journal of Cardiovascular Computed Tomography [in press]) of coronary CT angiograms in individuals undergoing pre-procedural assessment for transcatheter aortic valve replacement (n=36) demonstrate improved image quality of CCTA using SSF compared to CCTA not using SSF. Importantly, individuals in this study did not receive heart rate slowing agents (e.g., beta blockers), and diagnostic image quality was substantially improved. While not statistically powered on a per-patient basis, per-segment diagnostic accuracy of CCTA using SSF was superior to conventional CCTA. These results are complementary to those derived from internal testing at GE Healthcare wherein phantom work has demonstrated improved diagnostic performance using SSF compared to conventional image acquisitions.

Long-term Goal/Purpose: To demonstrate the incremental utility of SSF for individuals undergoing CCTA, with expected improvements in image quality and diagnostic accuracy. If the aims of this study are achieved, the use of SSF for effective temporal resolution improvement may obviate (or reduce) the need for CT hardware for improved temporal resolution.

ELIGIBILITY:
Inclusion Criteria:

1. Consenting adult patients ≥18 years of age;
2. Suspected but without known prior history of CAD
3. Not actively taking heart rate lowering agents at least 48 hours prior to study (e.g., AV nodal blockers such as beta blockers, calcium channel blockers or digoxin)
4. Glomerular filtration rate >60 ml/min
5. CCTA and ICA within 1 week of each other with no interscan event (e.g., myocardial infarction or coronary revascularization)

Exclusion Criteria:

1. Incomplete ICA or CCTA;
2. Known CAD (prior myocardial infarction, PCI, CABG)
3. Atrial Fibrillation
4. Abnormal Renal Function (GFR <60 ml/min)
5. Unwilling or unable to give consent
6. Non-cardiac illness with life expectancy <1 year
7. Concomitant participation in another clinical trial in which subject is subject to investigational drug or device
8. Pregnant women
9. Allergy to iodinated contrast agent
10. Contraindications to nitroglycerin
11. Systolic blood pressure ≤90 mm Hg
12. Contraindications to β blockers or nitroglycerin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consenting adult patients ≥18 years of age, Suspected but without known prior history of CAD, Not actively taking heart rate lowering agents at least 48 hours prior to study (e.g., AV nodal blockers such as beta blockers, calcium channel blockers or digoxin)
Sampling Method: Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2013-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy | 30 days
  To compare the per-patient, per-vessel and per-segment diagnostic accuracy of CCTA with SSF to conventional CCTA, as compared to invasive quantitative coronary angiography.
Diagnostic Interpretability | 30 days
  To compare the per-patient, per-vessel and per-segment diagnostic interpretability of CCTA with SSF to conventional CCTA, as compared to invasive quantitative coronary angiography.
Image quality | 30 day
  To compare the per-patient, per-vessel and per-segment quantitative image quality of CCTA with SSF to conventional CCTA, as compared to invasive quantitative coronary angiography.

SECONDARY OUTCOMES:
Upper threshold of heart rate | 1 day
  To determine the upper threshold of heart rate below which CCTA with SSF is most effective.
incremental & additive value | 1 day
  To determine the incremental & additive value of SSF to conventional CCTA for diagnostic accuracy / diagnostic interpretability / image quality.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (3):
  - MDDX, San Francisco, California
  - Walter Reed Medical Center, Bethesda, Maryland
  - Midwest Cardiology Associates, Independence, Missouri
- Diagnostico Maipu, San Isidro, Argentina
- University of British Columbia, Vancouver, British Columbia, Canada
- FACTS, Hyderabad, India
- Centro Cardiologico Monzino, Monzino, Italy